CLINICAL TRIAL: NCT06338215
Title: A Non-inferiority Randomized Trial Testing an Advice of Moderate Drinking Pattern Versus Advice on Abstention on Major Disease and Mortality
Brief Title: Advice of Moderate Drinking Pattern Versus Advice on Abstention on Major Disease and Mortality
Acronym: UNATI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNATI_2024; 101097681 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2024-03-13; First posted 2024-03-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-03

CONDITIONS: All Cause Mortality; Cardiovascular Diseases; Invasive Cancer; Liver Cirrhosis; Type 2 Diabetes; Depression; Dementia; Injury Traumatic; Tuberculosis; Infections
Keywords: Alcohol; Drinking Pattern; Abstention; Advice; Clinical Trial; Moderation; Mediterranean Alcohol Drinking Pattern
MeSH Terms: conditions — Cardiovascular Diseases; Liver Cirrhosis; Diabetes Mellitus, Type 2; Depression; Dementia; Wounds and Injuries; Tuberculosis; Infections | interventions — Ethanol

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderation (Experimental): Advice about alcohol intake following a Mediterranean Alcohol Drinking Pattern: Moderation (7 or less drinks/wk in women and 14 or less drinks/wk in men), avoidance of binge drinking, consumption of alcohol with meals and preference for red wine.
  Interventions: Behavioral: Moderate Alcohol Drinking Pattern; Behavioral: Abstention
- Abstention (Active Comparator): Advice on alcohol abstention.
  Interventions: Behavioral: Moderate Alcohol Drinking Pattern; Behavioral: Abstention

INTERVENTIONS:
Behavioral: Moderate Alcohol Drinking Pattern — Remotely Intensive intervention by specialized coaches (psychologists, dietitians, and other health professionals) to promote a behavior change on alcohol consumption. Repeated quarterly small group sessions and periodical personal interviews and educational videos, during up to 4 years with 1 contact every 3 months.
  Goals of intervention:
  1. moderate consumption (7 or less drinks/wk for women, 14 or less drinks/wk for men) of red wine (a drink=150 ml).
  2. always during meals
  3. spread out throughout the whole week, and
  4. avoidance of binge-drinking episodes. No participant will be invited to start or increase his/her alcohol intake.
Behavioral: Abstention — Remotely Intensive intervention by specialized coaches (psychologists, dietitians, and other health professionals) to promote a behavior change on alcohol consumption. Repeated quarterly small group sessions and periodical personal interviews and educational videos, during up to 4 years with 1 contact every 3 months.
  Goals of intervention:
  Abstention. Message of 0 alcohol.

SUMMARY:
The goal of this clinical trial is to test two advices on alcohol drinking in more than 10.000 Spanish adult drinkers (men of 50 or more years and women of 55 or more years).

The main question it aims to answer is to test the non-inferiority advice of a moderate alcohol drinking pattern on all-cause mortality and other chronic disease like cardiovascular disease, cancer or type 2 diabetes.

Participants will receive during 4 years an advice to drink alcohol following a Mediterranean Alcohol Drinking Pattern (MADP): consuming alcohol in moderation, avoidance of binge drinking and preference for red wine.

Researchers will compare those who will receive a MADP advice with those who will receive an advice on abstention to see if the advice on MADP is not inferior than the abstention advice to prevent all-cause mortality and other chronic diseases.

DETAILED DESCRIPTION:
Policymakers and clinicians are currently perplexed on how to reduce alcohol harms in drinkers, because of contradictory guidelines: abstention is proposed as the healthiest option by many health advocates, stating that "there is no safe level of alcohol intake"; but most nonrandomized studies found lower all-cause mortality and other beneficial outcomes in moderate drinkers than in abstainers among subjects >50 years. However, potential biases may compromise these latter studies, particularly when effects are null or moderate. A large pragmatic randomized controlled trial (RCT) of realistic advice aimed to change behaviour addressing clinical endpoints is long overdue. It will provide first-level evidence to confront the harms of one of the most widely used substances by humankind.

The European Research Council has funded, through an Advanced Research Grant (2023-2028) to the University of Navarra (Spain), as Host Institution, a 4-year non-inferiority RCT with more than 10,000 drinkers (men 50-70 years or women 55-75 years consuming 3 or more but 40 or less drinks/wk). The name of the trial is UNATI (University of Navarra Alumni Trialist Initiative).

At least ten thousand drinkers will be randomized in a 1:1 ratio to repeatedly (4 contacts/year) receive during 4 years two different advices:

1. abstention;
2. moderation (7 or less drinks/wk in women and 14 or less drinks/wk in men), avoidance of binge drinking, with preference for red wine consumed always with meals, and consumption spread out throughout the week, following the traditional Mediterranean Alcohol Drinking Pattern (MADP). Moderate consumption is hypothesized to be non-inferior. No initiation or increment in alcohol intake will be promoted.

The primary endpoint will be a global index of all-cause mortality, cardiovascular events, any invasive cancer, liver cirrhosis, type 2 diabetes, depression, dementia, injury requiring hospital admission or tuberculosis or other infections requiring hospitalization. As a secondary analysis, the most severe outcomes (mortality, invasive cancer, stroke, myocardial infarction, liver cirrhosis) will be considered independently with sufficient priority over less severe outcomes, using ad hoc methods.

The UNATI trial will provide for the first time an evidence-based answer to a question of the utmost interest in clinical medicine, given the high prevalence of moderate alcohol intake, and the current situation of equipoise with opposing views in the scientific community on the most sensible advice for moderate drinkers. The starting date for the project is December 1, 2023. The randomization of participants will start on June 2024.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 50-70 years, Women aged 55-75 years
* Drinkers of any alcoholic beverage initially consuming 3 or more but 40 or less drinks/wk
* Projected life expectancy more than 5 years (according to the judgment of their attending physician)
* Willing to receive advice during up to 4 years on how to improve their alcohol intake making it healthier

Exclusion Criteria:

1. Participants without smartphone or a computer (or tablet) with Internet connection.
2. Drinkers of less than 30 g of pure alcohol/wk or more than 400 g of pure alcohol/wk
3. Illiteracy, inability/unwillingness to give written consent or communicate with study staff, or inadequate abilities for the use of on-line technologies
4. Participants with any sever psychiatric condition or with a diagnosis of cognitive impairment or dementia.
5. Participants with liver cirrhosis or prior liver cancer.
6. Patients with a recent diagnosis of breast cancer (diagnosed in the last 10 years).
7. Patients under habitual use of high-dose medications that completely preclude any use of alcohol. Most of these patients will be already excluded by the second or fourth exclusion criteria.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison between groups of the incidence of a global Index of all-cause mortality and other alcohol-related diseases | From enrollment to the end of the intervention up to 4 years.
  Global index of all-cause mortality, cardiovascular events, any invasive cancer, liver cirrhosis, type 2 diabetes, depression, dementia, injury requiring hospital admission, tuberculosis or other infections requiring hospitalization evaluated from the information on clinical records.

SECONDARY OUTCOMES:
Comparison between groups of the incidence of the most severe outcomes | From enrollment to the end of the intervention up to 4 years
  The most severe outcomes (mortality, invasive cancer, stroke, myocardial infarction, liver cirrhosis) will be considered independently with sufficient priority over less sever outcomes, using ad hoc methods, using information on clinical records.

OTHER OUTCOMES:
Comparison between groups of invasive cancer incidence with extended follow-up | From the enrollment up to 10 or more years of follow-up
  The trial may not be long enough to observe effects on cancer endpoints. Therefore, a comparison between groups of cancer incidence endpoints after 10-year follow-up, assessed through the information on clinical records, will be included as an ancillary analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Martinez-Gonzalez, MD, MPH, PhD, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
The generated dataset (completely anonymized) will be made available to every proficient researcher who may present a relevant research proposal to the Steering Committee for further exploitation of the data upon all the usual legal precautions for the protection of individual data will be respected.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following the main article publication. Request out of these time frame can also be submitted.
Access Criteria: Researchers who provide a methodologically sound proposal approved by the UNATI Steering Committee.
URL: https://prevomnia.wixsite.com/proyectounati

REFERENCES:
- [Background] Martinez-Gonzalez MA. Should we remove wine from the Mediterranean diet?: a narrative review. Am J Clin Nutr. 2024 Feb;119(2):262-270. doi: 10.1016/j.ajcnut.2023.12.020. Epub 2023 Dec 28. PMID 38157987
- [Background] Martinez-Gonzalez MA, Hernandez Hernandez A. Effect of the Mediterranean diet in cardiovascular prevention. Rev Esp Cardiol (Engl Ed). 2024 Jul;77(7):574-582. doi: 10.1016/j.rec.2024.01.006. Epub 2024 Feb 7. English, Spanish. PMID 38336153
- [Background] Barberia-Latasa M, Bes-Rastrollo M, Perez-Araluce R, Martinez-Gonzalez MA, Gea A. Mediterranean Alcohol-Drinking Patterns and All-Cause Mortality in Women More Than 55 Years Old and Men More Than 50 Years Old in the "Seguimiento Universidad de Navarra" (SUN) Cohort. Nutrients. 2022 Dec 14;14(24):5310. doi: 10.3390/nu14245310. PMID 36558468